CLINICAL TRIAL: NCT06395610
Title: Open-label, Non-randomised, One-sequence Crossover Study to Investigate the Effect of Inhibition of CYP3A4/5 by Erythromycin on the Pharmacokinetics of CHF6001 in Healthy Subjects
Brief Title: Effect of Erythromycin on the Absorption, Metabolism and Elimination of CHF6001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLI-06001AA1-14; 2023-507300-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Drug-drug Interaction study; CYP3A4/5 inhibitor; CYP3A4/5 substrate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment R (Experimental): Single dose of CHF6001
  Interventions: Drug: CHF6001 DPI
- Treatment T (Experimental): Single dose of CHF6001 administered after repeated doses of oral Erythromycin
  Interventions: Drug: CHF6001 DPI; Drug: Erythromycin

INTERVENTIONS:
Drug: CHF6001 DPI — Single dose of CHF6001
Drug: Erythromycin — Repeated doses of oral Erythromycin
  Arms: Treatment T

SUMMARY:
The objective of this study is to investigate the effect of the interaction of Erythromycin (CYP3A4/5 moderate inhibitor) on the pharmacokinetic of CHF6001 (CYP3A4/5 substrate) in Healthy Volunteers.

DETAILED DESCRIPTION:
This clinical trial is a single centre, single dose Phase I study, with a non-randomized, open label, one sequence cross-over design.

A total of 24 healthy male and female are planned to be included. Participants will be dosed with CHF6001 before and during co-administration of Erythromycin and will act as their own control. The study will be run with a one-sequence crossover design, where all subjects will be treated with CHF6001 in the first treatment period and CHF6001+ Erythromycin in the second treatment period in order to avoid the need of a very long washout from the CYP3A4/5 inhibitor.

Standard safety assessments will be conducted during the Study, including safety blood and urine laboratory tests, vital signs, physical examinations, ECGs and observations of any adverse events. Blood samples will be also collected for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Healthy male and female subjects aged 18-55 years inclusive;
3. Ability to understand the study procedures, the risks involved and ability to be trained to use the inhalers correctly and to generate sufficient peak inspiratory flow (PIF) using the In Check device set as per NEXThaler® inhaler resistance;
4. Body mass index (BMI) between 18.0 and 35.0 kg/m2 extremes inclusive;
5. Non- or ex-smokers who smoked <5 pack-years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking >1 year prior to screening;
6. Good physical and mental status determined based on the medical history and a general clinical examination, at screening and before the first dosing;
7. Vital signs within normal limits at screening: diastolic blood pressure (DBP) 40-90 mmHg, systolic blood pressure (SBP) 90 140 mmHg (two measures performed after at least 5 min of resting; the mean value must be within the defined range);
8. A 12-lead digitalised electrocardiogram (ECG) considered as normal at screening: 40 bpm ≤ heart rate (HR) ≤110 bpm; 120 ms ≤ time interval between the P and R wave in the ECG (PR) ≤210 ms; 80 ms ≤ time interval between the Q and R and S wave in the ECG (QRS) ≤120 ms; Fridericia-corrected time interval between the Q and T wave in the ECG (QTcF) ≤450 ms for males and ≤470 ms for females;
9. Pulmonary function test within normal limits at screening: forced expiratory volume in the first second (FEV1) % predicted >80% and FEV1/forced vital capacity (FVC) ratio >0.70 (American Thoracic Society and European Respiratory Society [ATS/ERS] Task Force, 2019);
10. Female subjects:

    1. Women of childbearing potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method preferably with low user dependency (with exception of combined or progestogen-only hormonal contraception) from the signature of the informed consent and until the follow-up contact, or ii.WOCBP with non-fertile male partners: contraception is not required in this case;

       For the definition of WOCBP and of fertile men and the list of birth control methods with low user dependency, refer to Appendix 2 (or Section 4.1 of the Clinical Trial Facilitation Group guidance for more detailed information);

       Or
    2. Women of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. postmenopausal, or permanently sterile as per definitions given in Appendix 2). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per Investigator's request, postmenopausal status may be confirmed by follicle-stimulating hormone (FSH) levels (according to local laboratory ranges).

Exclusion Criteria:

1. Participation in another clinical trial where investigational drug was received, and last investigations were performed less than 8 weeks prior to screening;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic or psychiatric disorders, gastric surgery recently or in the past, and/or impaired Inclusion criteria: gastric motility that may interfere with successful completion of this protocol according to the Investigator's judgment;
3. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment;
4. Abnormal liver enzymes at screening (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >1.5x upper limit of normal [ULN]), bilirubin >1.5x ULN);
5. Subjects with history of breathing problems (e.g. history of asthma). Allergic asthma diagnosis in childhood (until 12 years old) is allowed;
6. Positive human immunodeficiency virus 1 or 2 (HIV1 or HIV2) serology at screening;
7. Positive results from the hepatitis serology which indicates acute or chronic hepatitis B (HB) or hepatitis C (HC) at screening (i.e. positive HB surface antigen [HBsAg], HB core antibody [IgM anti-HBc], HC antibody);
8. Blood donation or blood loss (equal or more than 450 mL) less than 8 weeks prior to screening or before the first dosing;
9. Positive urine test for cotinine at screening and before the first dosing;
10. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test at screening and before Treatment Period 1, Day -1;
11. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen evaluated at screening and before the first dosing;
12. Intake of non-permitted concomitant medication in the predefined period prior to screening or before the first dosing or the subject is expected to take non-permitted concomitant medication during the study;
13. Presence of any current infection, or previous infection that resolved less than 7 days prior to screening and before the first dosing;
14. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the trial;
15. Unsuitable arm veins for repeated venipuncture;
16. Heavy caffeine drinker (>5 cups or glasses of caffeinated beverages, e.g. coffee, tea, cola per day);
17. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test. Serum pregnancy test to be performed at screening and urine pregnancy test to be performed before the first dosing;
18. Subjects receiving treatment with any drug known to have a well defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, fluconazole, itraconazole, etc.) within the 3 months preceding the screening visit;
19. Subjects using e-cigarettes within 6 months before screening;
20. Positive test for coronavirus disease 2019 (COVID-19) (antibody test or nucleic acid test) within 14 days prior to screening and the associated complications/symptoms, which have not resolved within 14 days prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter (AUC0-t) | Over 96 hours after administration in blood
  Area under the curve from time 0 to the last quantifiable concentration (AUC0-t)
Pharmacokinetic parameter (Cmax) | Over 96 hours after administration in blood
  Maximum plasma concentration (Cmax) of CHF6001 without and with the concomitant administration of Erythromycin

SECONDARY OUTCOMES:
Pharmacokinetic parameter (AUC0-96) | Over 96 hours after administration in blood
  Area under plasma concentration from 0 to 96 hours (AUC0-96) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-∞) | Over 96 hours after administration in blood
  Area under curve extrapolated to infinity (AUC0-∞) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (tmax) | Over 96 hours after administration in blood
  Time to the maximum plasma concentration (tmax) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (CL/F) | Over 96 hours after administration in blood
  Apparent systemic clearance for CHF6001
Pharmacokinetic parameter (t1/2) | Over 96 hours after administration in blood
  Terminal elimination half-life (t1/2) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-t) | Over 96 hours after administration in blood
  Area under the plasma concentration versus time curve (AUC0-t) for CHF5956 and CHF6095
Pharmacokinetic parameter (Cmax) | Over 96 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF5956 and CHF6095

CONTACTS AND LOCATIONS:
Locations (1):
- MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No